CLINICAL TRIAL: NCT06983782
Title: CP-EXCEL: A Feasibility Randomised Controlled Trial of an Online Exercise Programme for Adults With Cerebral Palsy
Brief Title: A Feasibility Randomised Controlled Trial of an Online Exercise Programme for Adults With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC202501020
Record Dates: First submitted 2025-05-01; First posted 2025-05-21 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy; Exercise; Adults; Fitness
Keywords: Adults with cerebral palsy; Online exercise programme; physiotherapy
MeSH Terms: conditions — Cerebral Palsy; Motor Activity | interventions — Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Education (Experimental): Online exercise programme and educational material over 8 weeks.
  Interventions: Other: Exercise and education programme
- Placebo (Placebo Comparator): Educational materials over 8 weeks
  Interventions: Other: control group

INTERVENTIONS:
Other: Exercise and education programme — Participants will complete 8-week online exercise programme consisting of an online exercise class once per week. The exercises will target improving strength, balance and range of movement. In addition, participants will receive educational materials on exercise, nutrition, walking changes, fatigue, optimizing bone health, pain management, mental health, sleep and physical activity maintenance.
  Arms: Exercise and Education
Other: control group — The control group will receive educational materials over 8 weeks
  Arms: Placebo

SUMMARY:
Adults with cerebral palsy (CP) often face challenges in accessing exercise programmes that are appropriate for their needs. Barriers such as limited mobility, a lack of tailored options, and restricted access to physiotherapy services can make participation difficult. Exercise is important for improving physical health, mental well-being, and overall quality of life. However, many adults with CP do not have regular opportunities to take part in structured physical activity. This study aims to investigate whether an online exercise programme can serve as an effective and accessible alternative.

The main aim of the study is to assess the feasibility of delivering an online exercise programme for adults with CP. Key areas of focus will include demand, implementation, practicality, adaptability, acceptability, and potential benefits to physical, mental, and social well-being.

A total of 60 adults with CP will be recruited and randomly assigned to one of two groups (30 participants per group). One group will complete an 8-week online exercise and education programme. The second group will receive the same educational materials during the study and will be provided with information about the home exercise programme after the 8-week intervention period. Data will be collected on attendance, completion rates, engagement with exercises, and any reported adverse events. Health-related surveys will be completed before and after the programme to assess any changes. In addition, a selected group of participants from the intervention group will take part in interviews to provide feedback on their experiences.

Findings from this study may support the development of accessible, effective, and person-centred online exercise programmes for adults with CP. Results may help improve future programme design and contribute to better care and support for adults with CP in Ireland.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over with cerebral palsy (CP) residing on the island of Ireland.
* Individuals of any Gross Motor Function Classification System (GMFCS) level.
* Individuals with other associated impairments.
* People with mild-to-moderate intellectual disability who can access the online platform and follow study instructions, with or without support.

Exclusion Criteria:

* Individuals with severe intellectual disability where sufficient adaptations cannot be made.
* Adults with unstable medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Physical function | Duration of study 2 years
  Physical function will be measured using the PROMIS physical function- Short Form 10a scale.
Mobility | rolling recruitment over 1.2 years
  Mobility will be measured using the Functional mobility scale on a scale of 0-6.
Presence of Pain | Duration of study 2 years
  Pain will be assessed using a self-reported questionnaire, measured as Yes or No with description.

SECONDARY OUTCOMES:
Pain intensity | Duration of study 2 years
  Pain intensity will be measured using the PROMIS Pain intensity form
Pain quality | Duration of study 2 years
  Pain quality will be assessed using the PROMIS Neuropathic Pain Quality 5a and Nociceptive Pain Quality 5a scales, with total scores calculated for each to reflect the severity and type of pain experienced.
Pain interference | Duration of study 2 years
  Pain quality will be assessed using the PROMIS Pain interference Short Form-8a, with total scores calculated to reflect the quality of pain experienced.
Fatigue | Duration of study 2 years
  Fatigue will be assessed using the PROMIS Fatigue Short Form 13a (FACIT Fatigue) scale, with total scores calculated to reflect the severity of fatigue experienced by participants.
Sleep | Duration of study 2 years
  Sleep will be assessed using the PROMIS Sleep Disturbance Short Form 4a scale, with total scores reflecting the extent of sleep disturbance experienced by participants.
Self-efficacy | Duration of study 2 years
  Self-efficacy will be assessed using two PROMIS Short Form scales: the Self-Efficacy for Managing Chronic Conditions - Managing Daily Activities (Short Form 8a) and the Self-Efficacy for Managing Chronic Conditions - Managing Emotions. Total scores from each scale will reflect participants' confidence in managing daily activities and emotional responses related to their condition.
Depression | Duration of study 2 years
  Depression will be assessed using the PROMIS Emotional Distress - Depression Short Form 8a, with total scores reflecting the severity of depressive symptoms experienced by participants.
Participation | Duration of study 2 years
  Participation will be assessed using the PROMIS Ability to Participate in Social Roles and Activities Short Form 8a, with total scores indicating the extent to which participants are able to engage in social roles and daily activities.

OTHER OUTCOMES:
Practicality | Duration of study 2 years
  Practicality will be assessed by recording adverse events. Measured as Yes or No with description
Recruitment rate | Duration of study 2 years
  This will include recording the total number of people who responded to invitations or advertisements to participate in the study.
Fidelity to the intervention receipt | Duration of study 2 years
  Fidelity of intervention receipt will be measured by recording the number of sessions attended by participants in the intervention group throughout the study.
Fidelity of the intervention content | Duration of study 2 years
  Fidelity of intervention content will be assessed by self-reported completion of exercises, collected weekly from the intervention group and at follow-up from the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Ryan, PhD, Principal Investigator — Royal College of Surgeons in Ireland
Locations (1):
- Royal College of Surgeons in Ireland, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared due to concerns over participant confidentiality and the potential risk of re-identification.